CLINICAL TRIAL: NCT06973291
Title: A Phase 3, Randomized, Multicenter, Double-Blind Trial to Evaluate the Efficacy, Safety, and Tolerability of Zasocitinib (TAK-279) Compared to Deucravacitinib in Participants With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study Comparing Zasocitinib (TAK-279) With Deucravacitinib in Adults With Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-279-PsO-3004; 2024-512497-10-00 (EU CTIS Number); jRCT2011250014 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-05-08; First posted 2025-05-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
Keywords: Drug Therapy
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zasocitinib or Placebo (Experimental): Participants will receive zasocitinib or matching placebo tablet, orally, once daily (QD) up to Week 16.
  Interventions: Drug: Zasocitinib; Drug: Placebo to match zasocitinib
- Deucravacitinib or Placebo (Active Comparator): Participants will receive deucravacitinib 6 mg or matching placebo capsule, orally, QD up to Week 16.
  Interventions: Drug: Deucravacitinib; Drug: Placebo to match deucravacitinib

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib tablets.
  Other Names: TAK-279; NDI-034858
  Arms: Zasocitinib or Placebo
Drug: Deucravacitinib — Deucravacitinib capsules.
  Arms: Deucravacitinib or Placebo
Drug: Placebo to match zasocitinib — Zasocitinib matching placebo tablets.
  Arms: Zasocitinib or Placebo
Drug: Placebo to match deucravacitinib — Deucravacitinib matching placebo capsules.
  Arms: Deucravacitinib or Placebo

SUMMARY:
The main aim of this study is to assess whether zasocitinib works better than deucravacitinib in treating participants with moderate-to-severe plaque psoriasis.

Participants will take one tablet daily of either zasocitinib or a matching placebo, along with one capsule daily of either over-encapsulated deucravacitinib or a matching placebo, for a duration of 16 weeks.

Participants will be in the study for up to 25 weeks, which includes screening period of up to 35 days, a 16-week treatment period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a diagnosis of chronic plaque psoriasis for >=6 months prior to the screening visit.
2. Participant has stable plaque psoriasis, defined as no significant flare or change in morphology (as assessed by the investigator) in psoriasis, for >=6 months before screening.
3. Participant has moderate-to-severe plaque psoriasis, as defined by a PASI score >=12 and an sPGA score >=3, at screening and Day 1.
4. Participant has plaque psoriasis covering >=10 percent (%) of his or her total body surface area (BSA) at screening and Day 1.
5. Participant must be a candidate for phototherapy or systemic therapy.

Exclusion Criteria:

- Target Disease-Related Exclusions:

1. Participant has evidence of nonplaque psoriasis (erythrodermic, pustular, predominantly guttate psoriasis, predominantly inverse, or drug-induced psoriasis). If a participant meets criteria for inclusion based on typical plaque psoriasis presentation, a limited amount of inverse psoriasis is not exclusionary.
2. Participant requires systemic treatment, other than nonsteroidal anti-inflammatory drugs, during the trial period for an immune related disease (for example, inflammatory bowel disease).
3. Participant has a history of excessive sun exposure, has used tanning booths within 4 weeks prior to Day 1, or is not willing to minimize natural and artificial sunlight exposure during the trial period. Use of sunscreen products and protective apparel is recommended when sun exposure cannot be avoided.
4. Participant has concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the trial assessments.

   Recent/Concurrent Infectious Disease Exclusions:
5. Tuberculosis (TB):

   1. Participant has history of active TB infection, regardless of treatment status.
   2. Participant has signs or symptoms of active TB (including, but not limited to, chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator.
   3. Participant has evidence of latent TB infection (LTBI) as evidenced by a positive QuantiFERON-TB Gold (QFT) result OR 2 indeterminate QFT results, and participant does not have documentation of appropriate LTBI prophylaxis or is not able or not willing to initiate appropriate LTBI prophylaxis.
   4. Participant has had any imaging trial during or 6 months prior to screening, including x-ray, chest computed tomography, Magnetic Resonance Imaging (MRI), or other chest imaging suggesting evidence of current active or a history of active TB. X-ray is required for all participants regardless of QFT results unless the participant has had normal chest imaging in the 6 months prior to screening.
6. Herpes infections:

   1. Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1.
   2. Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
7. Nonherpetic viral diseases:

   1. Participant has presence of Hepatitis C Virus (HCV) antibody and a positive confirmatory test result for HCV ribonucleic Acid (RNA) (nucleic acid test or Polymerase Chain Reaction [PCR]).
   2. Participant has presence of positive Hepatitis B Surface Antigen (HBsAg+), or indeterminate HBsAg, presence of HBV deoxyribonucleic Acid (DNA) (regardless of serology), or positive anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody (Hepatitis B Core Antibody [HBcAb] positive and Hepatitis B Surface Antibody [HBsAb] negative).
   3. Participant has positive results for Human Immunodeficiency Virus (HIV) by serology, regardless of viral load.
8. Other infectious diseases:

   1. Participant has a history of active infection or febrile illness within 7 days prior to Day 1, as assessed by the investigator.
   2. Participant has history of symptoms suggestive of systemic or invasive infection within 30 days prior to Day 1.
   3. Participant has history of bacterial, viral, or fungal infection that required hospitalization or treatment with intravenous antimicrobial therapy within 8 weeks prior to Day 1 or oral antimicrobial therapy within 30 days prior to Day 1.
   4. Participant has a history of chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial onychomycosis).
   5. Participant has a history of an infected joint prosthesis, unless that prosthesis has been removed or replaced at least 60 days prior to Day 1.
   6. Participant has a history of opportunistic infections (for example, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   7. Participant had a bacterial infection within 60 days prior to Day 1 for which he or she did not receive treatment.

      * Noninfectious Disorders Exclusions:
9. Participant has any clinically significant medical condition, evidence of an unstable clinical condition (for example, cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or immunologic), or vital signs/physical/laboratory/Electrocardiogram (ECG) abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of trial results. These include but are not limited to:

   1. Participant has a history of known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency, splenectomy.
   2. Participant had a major surgery within 60 days prior to Day 1 or has a major surgery planned during the trial.
   3. Participant has unstable, poorly controlled, or severe hypertension at screening, confirmed by 2 repeat assessments.
   4. Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association criteria.
   5. Participant has a history of cancer or lymphoproliferative disease, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
   6. For participants with asthma, chronic obstructive pulmonary disease, or other pulmonary illnesses, participant has been hospitalized in the past 3 months, has ever required intubation for treatment, currently requires oral corticosteroids, or has required more than 1 course of oral corticosteroids within 6 months prior to Day 1.
   7. Participant has any of the following cardiovascular disease history:

      * A new diagnosis of atrial fibrillation or an episode of atrial fibrillation with rapid ventricular response or other dysrhythmia, nonacute cardiac hospitalization (for example, pacemaker implantation), pulmonary embolism, or deep venous thrombosis within the past 6 months prior to screening.
      * Any history of cerebrovascular event, myocardial infarction, coronary stenting, or aorto-coronary bypass surgery. If, however, the investigator determines there are no suitable treatment alternatives available for the participant and it has been at least 6 months since the occurrence of any such event, the participant may enroll.
   8. Participant has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the trial, in the opinion of the investigator.
   9. Participant has significant/uncontrolled psychiatric illness, in the opinion of the investigator.
   10. Participant has a history of clinically significant drug or alcohol abuse within 12 months prior to Day 1.

       * Prohibited Psoriasis Treatments Exclusions:

   For the below prohibited psoriasis treatments, the washout period prior to Day 1 is within the time frame indicated or 5 half-lives, whichever is longer, regardless of whether they are prescribed for psoriasis or another condition:
10. Participant has received any of the following biologics or biosimilar versions within the time frame indicated:

    1. Antibodies to interleukin (IL)-12/-23, IL-17, or IL-23 (for example, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab) within 6 months prior to Day 1.
    2. Tumor Necrosis Factor (TNF) inhibitor(s) (for example, etanercept, adalimumab, infliximab, or certolizumab) within 2 months prior to Day 1.
    3. Agents that modulate integrin pathways to impact lymphocyte trafficking (for example, natalizumab) or agents that modulate B cells or T cells (for example, alemtuzumab, abatacept, or visilizumab) within 3 months prior to Day 1.
    4. Rituximab or other immune cell-depleting therapy within 6 months prior to Day 1.
11. Participant has used medicated shampoo and/or body wash, including formulations containing but not limited to salicylic acid, corticosteroids, coal tar, vitamin D3 analogues, or other compounds used for the management of psoriasis within 2 weeks prior to Day 1.
12. Participant has used any topical medication that could affect psoriasis presentation (including but not limited to corticosteroids, salicylic acid, urea, alpha- or beta-hydroxy acids, anthralin, retinoids, vitamin D analogues [such as calcipotriol], methoxsalen, trimethylpsoralen, calcineurin inhibitors [for example, tacrolimus], tapinarof, roflumilast, Janus kinase (JAK) inhibitors, or tar) within 2 weeks prior to Day 1.
13. Participant has used any systemic nonbiologic treatment that could affect psoriasis presentation (including oral, intravenous, intramuscular, intra-articular, intrathecal, or intralesional corticosteroids; oral retinoids; immunosuppressive/immunomodulating medication; methotrexate; azathioprine; 6-thioguanidine; mercaptopurine; mycophenolate mofetil; hydroxyurea; cyclosporine; 1,25-dihydroxyvitamin D3 analogues; psoralens; sulfasalazine; fumaric acid derivatives; JAK inhibitors; apremilast) within 4 weeks prior to Day 1, or 5 half-lives, whichever is longer. Note: Intranasal corticosteroids, inhaled corticosteroids, and eye and ear drops containing corticosteroids are permitted.
14. Participant has used leflunomide within 6 months prior to Day 1.
15. Participant has received phototherapy (including Ultraviolet B [UV B], Psoralen plus Ultraviolet A [PUVA], tanning beds, therapeutic sunbathing) or excimer laser within 4 weeks prior to Day 1.
16. Participant has used botanical preparations (for example, herbal supplements or traditional medicines, including traditional Chinese medicines derived from plants, minerals, or animals) intended to treat psoriasis or other immunological diseases within 4 weeks prior to Day 1.
17. Participant is currently being treated with oral antihistamines for any reason, with the exception of oral antihistamines that are administered at a stable dose for at least 4 weeks prior to Day 1. Note: Additional treatment with oral antihistamines may be permitted after discussion with the medical monitor.
18. Participant has any previous exposure to zasocitinib (also known as TAK-279 or NDI 034858) or other Tyrosine Kinase 2 (TYK2) inhibitors (including deucravacitinib), or participated in any trial that included a TYK2 inhibitor (for example, deucravacitinib, VTX958, GLPG3667, et cetera), unless participant has documentation of posttrial unblinding that confirms the participant did not receive a TYK2 inhibitor.

    - Other Prohibited Concomitant Medications Exclusions: For the below prohibited concomitant medications, where applicable, the washout period prior to Day 1 is within the time frame indicated or 5 half-lives, whichever is longer.
19. Participant has received lithium, antimalarials, or intramuscular gold therapy within 4 weeks prior to Day 1.
20. Participant is currently being treated with strong or moderate Cytochrome P450 3A4 (CYP3A4) inhibitors (such as itraconazole) or strong or moderate CYP3A4 inducers (such as rifampin, carbamazepine, or phenytoin), or has received strong or moderate CYP3A4 inhibitors or strong or moderate CYP3A4 inducers within 4 weeks or 5 half-lives of the inducer or inhibitor, whichever is longer, prior to Day 1, or is anticipated to require treatment with strong or moderate CYP3A4 inducers or inhibitors during the trial period.

    Note: This includes consumption of food or beverages containing grapefruit and/or Seville oranges within 1 week of Day 1. Participants must be counseled to avoid food or beverages containing grapefruit and/or Seville oranges for the duration of the trial.
21. Participant has received any live-attenuated vaccine within 60 days prior to Day 1 or plans to receive a live-attenuated vaccine during the trial and up to 4 weeks after the last trial intervention administration.

    Note: Non-live-attenuated vaccines or boosters for Coronavirus Disease 2019 (COVID-19) or influenza are permitted during the trial.
22. Participant received an investigational antibody or biologic therapy within 6 months prior to Day 1.
23. Participant received an investigational oral therapy within 3 months prior to Day 1.
24. Participant is currently receiving a nonbiological trial intervention or device or has received one within 4 weeks prior to Day 1.
25. Participant is currently enrolled in a clinical trial or anticipates enrollment in a clinical trial during the course of the trial.

    - Laboratory/Physical Exclusions:
26. Participant has any of the following laboratory values at the screening visit:

    1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values greater than (˃)3*upper limit of normal (ULN).
    2. Total Bilirubin (Tbili) (unconjugated and/or conjugated) ˃1.5*ULN.
    3. Hemoglobin less than (<) 9.0 grams per deciliter (g/dL) (<90.0 grams per liter [g/L]).
    4. Absolute white blood cell (WBC) count <3.0*109/liters (L) (<3000 per cubic millimeter [/mm3]).
    5. Absolute neutrophil count of <1.0*109/L (<1000/mm3).
    6. Absolute lymphocytes count of <0.5*109/L (<500/mm3).
    7. Platelet count <100*109/L (<100,000/mm3).
    8. Thyroid-stimulating hormone outside the normal reference range AND free T4 or T3 outside the normal reference range.
    9. Estimated creatinine clearance <45 milliliters per minute (mL/min) based on the Cockcroft-Gault calculation.
    10. Creatine phosphokinase (CPK) > ULN. CPK may be repeated once; if repeat value is Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or lower (or <=2.5*ULN) and no higher than the initial value, participant remains eligible. Investigators should assess the participant for modulating factors, including concomitant medications or vigorous exercise, that may affect CPK levels.
27. Participant has any other significant laboratory abnormalities that, in the opinion of the investigator, might place the participant at unacceptable risk for participation in this trial.
28. Participant does not tolerate venipuncture or inability to be venipunctured.

    - Allergies and Adverse Drug Reactions Exclusions:
29. Participant has history of significant drug allergy (such as anaphylaxis).
30. Participant has a known or suspected allergy to zasocitinib or deucravacitinib or any of their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI)-100 at Week 16 | At Week 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (less than or equal to [<=] 3 representing mild disease, greater than or equal to [>=3] to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100 percentage (%) improvement in PASI score relative to baseline PASI score will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving PASI-90 at Weeks 4, 8, 12, and 16 | At Weeks 4, 8, 12, and 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (<= 3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI <=2 Response at Weeks 4, 8, 12, and 16 | At Weeks 4, 8, 12, and 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (<= 3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Percentage of participants achieving PASI <=2 at Weeks 4, 8, 12, and 16 will be reported.
Percentage of Participants Achieving Static Physician's Global Assessment (sPGA) of Clear (0) at Weeks 4, 8, 12, and 16 | At Weeks 4, 8, 12, and 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants Achieving PASI-100 at Weeks 4, 8, and 12 | At Weeks 4, 8, and 12
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (<= 3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-75 at Weeks 4, 8, 12, and 16 | At Weeks 4, 8, 12, and 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving sPGA of Clear (0) or Almost Clear (1) at Weeks 4, 8, 12, and 16 | At Weeks 4, 8, 12, and 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Change From Baseline in PASI Score at Weeks 4, 8, 12, and 16 | Baseline, Weeks 4, 8, 12, and 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (<= 3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Change from baseline will be calculated as post-baseline value minus baseline value.
Percent Change From Baseline in PASI score at Weeks 4, 8, 12, and 16 | Baseline, Weeks 4, 8, 12, and 16
  PASI is a measure of the average erythema, induration/infiltration, and desquamation/scaling of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72 (<= 3 representing mild disease, >=3 to 15 representing moderate disease, and >=15 indicating severe disease) with higher PASI scores denoting more severe disease activity. Percent change from baseline will be calculated as post-baseline value minus baseline value multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (113):
- United States (31):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Zenith Research, Inc., Beverly Hills, California
  - First OC Dermatology Research Inc., Fountain Valley, California
  - UNISON Clinical Trials (Shahram Jacobs md inc.), Sherman Oaks, California
  - Central Connecticut Dermatology, PLLC, Cromwell, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Direct Helpers Research Center, Hialeah, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Endeavor Health Clinical Trials, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Markowitz Medical PLLC dba OptiSkin Medical, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Bexley Dermatology Research - Probity - PPDS, Bexley, Ohio
  - Apex Clinical Research Center, LLC - Canton, Canton, Ohio
  - Apex Clinical Research Center, LLC - Mayfield Heights, Mayfield Heights, Ohio
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - The University of Texas Health Science Center at Houston (UTHSC-H), Bellaire, Texas
  - Reveal Research Institute, Dallas, Texas
  - San Antonio, San Antonio, Texas
  - Texas Dermatology and Laser Specialists-San Antonio, San Antonio, Texas
  - Houston Center for Clinical Research, LLC, Sugar Land, Texas
- Bulgaria (10):
  - Medical Centre Femiclinic EOOD, Sofia, Dianabad District
  - Medical Center Unimed EOOD-Sevlievo, Sevlievo, Gabrovo
  - Medical Center Asklepii OOD, Dupnitsa, Kyustendil
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - Medical Center Hera EOOD-Sofia, Sofia, Sofia-Grad
  - Diagnostic Consultative Center XXVIII - Sofia - EOOD, Sofia, Sofia-Grad
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Diagnostic Consultative Center Sveti Georgi EOOD, Haskovo
  - Medical Center Medconsult Pleven - Lovech Branch, Lovech
- Canada (18):
  - Beacon Dermatology - Probity, Calgary, Alberta
  - VIDA Dermatology - Probity, Edmonton, Alberta
  - Enverus Medical Research - Probity, Surrey, British Columbia
  - Dr Chih-Ho Hong Medical Inc, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Brunswick Dermatology Centre - Probity, Fredericton, New Brunswick
  - Lima's Excellence In Allergy And Dermatology Research (Leader) Inc. - Probity, Hamilton, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Lynderm Research Inc - Probity, Markham, Ontario
  - North Bay Dermatology Center - Probity, North Bay, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre For Dermatology, Richmond Hill, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Siena Medical Research Corporation, Montreal, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec
- Czechia (8):
  - Nemocnice AGEL Novy Jicin a.s, Nový Jičín, Moravskoslezský kraj
  - CCR Ostrava s.r.o., Ostrava, Moravskoslezský kraj
  - Dermskin s.r.o, Olomouc, Olomoucký kraj
  - Pratia Brno s.r.o. - PRATIA - PPDS, Brno, South Moravian
  - Pratia Pardubice, Pardubice
  - CLINTRIAL s.r.o., Prague
  - Prof. MUDr. Petr Arenberger, DrSc. - CRC - PPDS, Prague
  - Praglandia s.r.o., Prague
- France (4):
  - Office of Mireille Ruer-Mulard, MD, Martigues, Paca
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Hopital Charles Nicolle-1 Rue de Germont, Rouen
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
- Japan (15):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Hino Dermatology Clinic, Fukutsu-shi, Fukuoka
  - JR Sapporo Hospital, Sapporo, Hokkaido
  - Investigational Product department, Sapporo, Hokkaido
  - Nippon Life Hospital, Osaka, Osaka
  - Investigational Product department Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Seikoukai Omi Medical Center, Kusatsu-shi, Shiga
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - Medical Corporation Jitai-kai Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo-to
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
  - Ohyama Dermatology Clinic, Kumamoto
- Latvia (7):
  - Semigallia, Kuldīga
  - Health Center 4, Center of Diagnostics, Riga
  - Health Center 4, Clinic of Dermatology, Riga
  - Riga 1st Hospital, Riga
  - Aesthetic dermatology clinic of prof. J. Kisis, Riga
  - Veseliba un estetika Ltd., Riga
  - Outpatient Clinic Adoria, Riga
- Poland (20):
  - DermoDent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski, s.c., Osielsko, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Swietokrzyski, Lower Silesian Voivodeship
  - Cityclinic Przychodnia lekarsko psychologiczna Matusiak sp.p, Wroclaw, Lower Silesian Voivodeship
  - Centrum Columbus, Wroclaw, Lower Silesian Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Dorota Krasowska, Lublin, Lublin Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park Sp. z o.o. sp. k. | Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - ETG Warszawa - PPDS, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - ClinicMed Daniluk, Nowak Spolka Komandytowa, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych Pi-house Sp. Z O. O., Gdansk, Pomeranian Voivodeship
  - Ambulatorium Sp. z o.o. | Elblag, Poland, Elblag, Warmian-Masurian Voivodeship
  - NZOZ Holsamed-Oddział Libero, Katowice
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Centrum Terapii Współczesnej J.M. Jasnorzewska S.K.A., Lodz, Łódź Voivodeship
  - Dermoklinika-Centrum Medyczne s.c, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/find-a-trial?idFilter=TAK-279-PsO-3004